CLINICAL TRIAL: NCT03649711
Title: A Mechanistic Study in Patients With Non-Dialysis Chronic Kidney Disease to Investigate Altered Platelet Response to Antiplatelet Therapy (CKD-Platelet Study)
Brief Title: Chronic Kidney Disease (CKD) Platelet Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Arkansas (Other)
Collaborators: American Society of Nephrology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 227997; 1241997 (Other: Central Arkansas Veterans Affairs Hospital)
Record Dates: First submitted 2018-08-21; First posted 2018-08-28 (Actual); Results first posted 2022-12-29 (Actual); Last update posted 2022-12-29 (Actual); Status verified 2022-08

CONDITIONS: Chronic Kidney Diseases; Heart Attack; Stroke, Ischemic
Keywords: P2Y12 inhibitors; Platelet aggregation; ticagrelor; clopidogrel; chronic kidney disease
MeSH Terms: conditions — Renal Insufficiency, Chronic; Myocardial Infarction; Ischemic Stroke | interventions — Ticagrelor; Clopidogrel; Aspirin

STUDY DESIGN:
Intervention Model Description: CKD participants will be double-blind randomized in these two arms:
  Arm 1 - Ticagrelor, 90 mg twice daily (one pill in the morning and one pill in the evening) + Aspirin 81 mg/day. Ticagrelor is the test treatment.
  Arm 2 - Clopidogrel, 75 mg/day in the morning and a matching placebo in the evening + Aspirin 81 mg/day. Clopidogrel is the reference treatment.
  Arm 3: Control with normal kidney function will be recruited after matching for age and diabetes status to the Arm 1 participants. Participants will be asked to take Ticagrelor, 90 mg twice daily (one pill in the morning and one pill in the evening) and aspirin 81 mg/day. Open label treatment.
  All participants are required to take the oral treatment for a total of two weeks.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: CKD participants will be randomly assigned into one of the 2 study groups: ticagrelor (90 mg) one pill in the morning and one pill in the evening, or, clopidogrel (75 mg) one pill in the morning + placebo one pill in the evening. Placebo looks like the study drug but has no medicine in it. Neither participant nor the study personnel will know about allocation. The study drugs will look the same, except aspirin pill which will be dispensed to everyone in an open label manner.
  There is no masking for control with normal kidney function. Participants will be asked to take open label ticagrelor, 90 mg twice daily (one pill in the morning and one pill in the evening) and aspirin 81 mg/day.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- CKD-Ticagrelor (Experimental): Ticagrelor 90 mg twice daily (double blind, random assignment) + aspirin 81 mg/d
  Interventions: Drug: Ticagrelor 90mg; Drug: Aspirin 81 mg
- CKD-Clopidogrel (Active Comparator): Clopidogrel 75 mg/day in the morning and a matching placebo in the evening to conceal frequency (double blind, random assignment) + aspirin 81 mg/d
  Interventions: Drug: Clopidogrel 75mg; Drug: Aspirin 81 mg
- Control-ticagrelor (Active Comparator): Open label ticagrelor, 90 mg twice daily + aspirin 81 mg/d
  Interventions: Drug: Ticagrelor 90mg; Drug: Aspirin 81 mg

INTERVENTIONS:
Drug: Ticagrelor 90mg — Ticagrelor Pill
  Other Names: Brilinta
  Arms: CKD-Ticagrelor; Control-ticagrelor
Drug: Clopidogrel 75mg — Clopidogrel Pill and a matching placebo to conceal frequency
  Other Names: Plavix
  Arms: CKD-Clopidogrel
Drug: Aspirin 81 mg — Aspirin Pill
  Other Names: baby aspirin

SUMMARY:
This study evaluates how aspirin, clopidogrel and ticagrelor work in people with chronic kidney disease (CKD) compared to people with normal kidneys. In the first part of the study, half of CKD participants will be randomly assigned to ticagrelor and aspirin, while the other half will be assigned to clopidogrel and aspirin in a blinded fashion. The treatment duration will be two weeks. After recruiting CKD participants the investigator will recruit controls with normal kidney function that will receive only ticagrelor and aspirin for two weeks.

DETAILED DESCRIPTION:
It is known that people with chronic kidney disease (CKD) are at higher risk to have heart and blood vessel problems like heart attack and stroke compared to people that do not have kidney problems. Aspirin, clopidogrel and ticagrelor prevent blood clots building up in the vessels. If a blood clot is present in one vessel, it could stop oxygen carrying blood to get to a specific organ, and that could cause problems like heart attack or stroke. There is very little knowledge about the way this group of medicines works in people with chronic kidney disease as well as it works in individuals with normal kidney function.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females, aged 18-91 years
2. Ability to understand and sign informed consent after the nature of the study has been fully explained
3. CKD participants: Non-dialysis CKD patients: Presence of CKD with an estimated GFR of <30 mL/min/1.73 m2 for a period of ≥3 months, as defined by the National Kidney Foundation (NKF) and determined with the CKD-EPI creatinine-based formula
4. Controls with normal kidney function: participants with an estimated GFR >90 mL/min/1.73 m2 as determined by the CKD-EPI creatinine-based formula and a urine albumin-to-creatinine ratio <30 mg/g as defined by the National Kidney Foundation

Exclusion Criteria:

* No healthcare power of attorney to sign informed consent
* Unwillingness or inability to participate in the protocol or comply with any of its components.
* Subjects unable or unwilling to stop taking:

  * Aspirin and other antithrombotic agents, like cilostazol, ranolazine, aggrenox, prasugrel, warfarin, xarelto, pradaxa, eliquis.
  * Glycoprotein IIb/IIIa antagonist (abciximab-ReoPro, eptifibatide-Integrilin, tirofiban-Aggrastal)
  * NSAIDs and PPIs
  * Fish oil, Vitamin E and herbal supplements
* Acute kidney injury superimposed on CKD
* Kidney transplant or any other solid organ transplant recipient
* End-stage kidney disease on maintenance dialysis (peritoneal or hemodialysis)
* Nephrotic syndrome defined as nephrotic range proteinuria, hypoalbuminemia, hyperlipidemia and generalized edema
* Recent hospitalization or surgery <3 months
* Acute coronary or cerebrovascular event in the last 12 months
* Blood dyscrasias, active bleeding, or bleeding diathesis
* Gastrointestinal bleeding in the last 6 months
* Recent treatment (<30 days) with a glycoprotein IIb/IIIa antagonist (Integrelin).
* Hematocrit <25%, white blood cell count >20,000/μL, or platelet count <50,000/μL
* Any active malignancy or liver disease.
* Pregnancy
* Positive urine pregnancy test in a woman of childbearing potential prior to study entry. A female of childbearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

  * Has not undergone a hysterectomy or bilateral oophorectomy; or
  * Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).
* Patients must not be nursing due to the potential for congenital abnormalities and the potential of this regimen to harm nursing infants.

Ages: 18 Years to 91 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2021-09-02 (Actual); Study Completion 2021-09-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jain Nishank, MD, Principal Investigator — University of Arkansas for Medical
Locations (2):
- United States (2):
  - Central Arkansas Veterans Affairs Hospital, Little Rock, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas

IPD SHARING:
Plan to Share IPD: Yes
De-identified data for all primary and secondary outcome measures will be uploaded on clinicaltrials.gov website.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 2 years after study closure indefinitely

REFERENCES:
- [Derived] Jain N, Corken A, Arthur JM, Ware J, Arulprakash N, Dai J, Phadnis MA, Davis O, Rahmatallah Y, Mehta JL, Hedayati SS, Smyth S. Ticagrelor inhibits platelet aggregation and reduces inflammatory burden more than clopidogrel in patients with stages 4 or 5 chronic kidney disease. Vascul Pharmacol. 2023 Feb;148:107143. doi: 10.1016/j.vph.2023.107143. Epub 2023 Jan 20. PMID 36682595
- [Derived] Natale P, Palmer SC, Saglimbene VM, Ruospo M, Razavian M, Craig JC, Jardine MJ, Webster AC, Strippoli GF. Antiplatelet agents for chronic kidney disease. Cochrane Database Syst Rev. 2022 Feb 28;2(2):CD008834. doi: 10.1002/14651858.CD008834.pub4. PMID 35224730
- See also: publication — https://kidney360.asnjournals.org/content/early/2022/10/26/KID.0005532022

RESULTS

PARTICIPANT FLOW:
Recruitment Details: CKD recruitment. 50 patients signed consent and were randomized. Of those randomized, 1 received kidney transplant and 1 allergic reaction to clopidogrel and did not complete the study visits. 48 patients completed study visits.
  Non-CKD control recruitment: 26 signed consent and completed study visits.
Pre-assignment Details: Goal 48 CKD who complete visits; we ended up consenting and randomizing 50 CKD patients.
  Enrolled 26 to achieve goal. actual enrollment 50+26 = 76
Groups:
- Experimental: CKD-Ticagrelor: Ticagrelor 90 mg twice daily (double blind, random assignment) + aspirin 81mg/d
- Arm: Active Comparator: CKD-Clopidogrel: Clopidogrel 75mg/day in the morning and a matching placebo in the evening to conceal frequency (double blind, random assignment) + aspirin 81 mg/d
- Non-CKD Control Arm: Active Comparator: Control-ticagrelor: Open label ticagrelor, 90 mg twice daily + aspirin 81 mg/d in subjects recruited without CKD
Period: Overall Study
Arm/Group | Experimental: CKD-Ticagrelor | Arm: Active Comparator: CKD-Clopidogrel | Non-CKD Control Arm: Active Comparator: Control-ticagrelor
Started | 26 | 24 | 26
Completed | 25 | 23 | 26
Not Completed | 1 | 1 | 0
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Kidney Transplant | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Experimental: CKD-Ticagrelor: Ticagrelor 90mg Twice daily (double blind, random assignment) + aspirin 81 mg/d
- Active Comparator: CKD-Clopidogrel: Clpidogrel 75 mg/day in the morning and a matching placebo in the evening to conceal frequency (double blind, random assignment) aspirin 81 mg/d
- Non-CKD Control Arm - Active Comparator: Control-ticagrelor: Open label ticagrelor, 90 mg twice daily + aspirin 81 mg/d in subjects without CKD
- Total: Total of all reporting groups
Arm/Group | Experimental: CKD-Ticagrelor | Active Comparator: CKD-Clopidogrel | Non-CKD Control Arm - Active Comparator: Control-ticagrelor | Total
Number analyzed (Participants) | 25 | 23 | 26 | 74
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.2 (11.5) | 52.2 (15.1) | 48.0 (15.2) | 52.2 (15.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 16 | 42
  Male | 12 | 10 | 10 | 32
Race/Ethnicity, Customized [Number; unit: participants]
  African American | 13 | 13 | 3 | 29
  Caucasian | 11 | 9 | 21 | 41
  Hispanics | 1 | 0 | 2 | 3
  Asian | 0 | 1 | 0 | 1
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 34.5 (8.6) | 32.5 (9.1) | 31.2 (7.0) | 33.5 (8.8)
Diabetes mellitus, n (%) [Count of Participants; unit: Participants] | 17 | 14 | 0 | 31
Statin use, n (%) [Count of Participants; unit: Participants] | 15 | 14 | 4 | 33
Baseline use of aspirin, n (%) [Count of Participants; unit: Participants] | 10 | 7 | 3 | 20
Serum creatinine [Mean (Standard Deviation); unit: mg/dl] | 4.2 (1.9) | 4.3 (1.8) | 0.9 (0.1) | 4.2 (1.9)
eGFR [Mean (Standard Deviation); unit: mL/min/1.73 m^2] | 16.7 (6.5) | 16.4 (5.7) | 89.6 (13.2) | 16.5 (6.0)
Urine albumin-to-creatinine ratio [Median (Inter-Quartile Range); unit: mg/g of creatinine] | 1,039.0 [715.6 to 2,382.5] | 2,400.0 [519.7 to 4,243.0] | 0 [0 to 0] | 1,229.4 [638.0 to 3,329.0]
Hemoglobin [Mean (Standard Deviation); unit: g/dl] | 11.1 (1.8) | 11.1 (1.9) | 13.5 (1.3) | 13.5 (1.3)
White blood cell count [Mean (Standard Deviation); unit: 1000 cells per µL] | 7.7 (2.4) | 7.5 (2.4) | 6.2 (1.6) | 7.6 (2.4)
Platelet count [Median (Standard Deviation); unit: 1000 cells per µL] | 243.07 (71.1) | 229.9 (49.7) | 266.5 (57.9) | 236.7 (61.5)
Percent of Hemoglobin A1c [Mean (Standard Deviation); unit: percentage of hemoglobin] | 6.9 (1.6) | 7.0 (1.9) | 5.3 (0.4) | 6.9 (1.6)

OUTCOME MEASURES:

1. Primary Outcome: ADP Induced Platelet Aggregation
Description: We will use summary statistics to describe the distribution of the data. Post-treatment ADP-induced WBPA value in ohms (Ω) will be the primary outcome variable. We will use an analysis of covariance (ANCOVA) model to compare the treatment effects of ticagrelor vs. clopidogrel in CKD patients because this approach has higher statistical power than other methods to analyze drug effects. T
Time Frame: 2 weeks
Population: CKD groups were analyzed between randomized arms using ANCOVA. CK-ticagrelor arm was compared to control ticagrelor arm using Wilcoxon rank sum test.
Measure: Median (Inter-Quartile Range); unit: ohms
Arm/Group | CKD-Ticagrelor | CKD-Clopidogrel | Control-ticagrelor
Number analyzed (Participants) | 25 | 23 | 26
ohms | 0 [0 to 2] | 6 [1 to 10.5] | 1 [0 to 3]
Statistical Analysis 1: Comparison: CKD-Ticagrelor vs CKD-Clopidogrel; Test type: Other — Post treatment values were compared using ANCOVA; p = 0.002, ANCOVA
Statistical Analysis 2: Comparison: CKD-Ticagrelor vs Control-ticagrelor; mean changes in values were compared by Wilcoxon rank sum test adjusted for multiple comparisons (Bonferonni method) between CKD-ticagrelor arm, and the non-CKD controls; Test type: Other; p = 0.18, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Platelet Surface P-selectin Expression
Description: Platelet surface P-selectin expression was measured using flow cytometry before and after treatment.
Time Frame: 2 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Fluorescence intensity
Arm/Group | CKD-Ticagrelor | CKD-Clopidogrel | Control-ticagrelor
Number analyzed (Participants) | 25 | 23 | 26
Fluorescence intensity | 1002.5 [758.5 to 1149.5] | 1037.5 [848.5 to 1262.75] | 1052 [810 to 1279]
Statistical Analysis 1: Comparison: CKD-Ticagrelor vs CKD-Clopidogrel; CKD groups randomized were compared for post treatment values; Test type: Other; p = 0.22, ANCOVA

ADVERSE EVENTS:
Time Frame: Adverse events reported during the 2 weeks of treatment from baseline visit to the final visit
Groups:
- Arm: Active Comparator: Control-ticagrelor: Open label ticagrelor, 90 mg twice daily + aspirin 81 mg/d
Arm/Group | Experimental: CKD-Ticagrelor | Arm: Active Comparator: CKD-Clopidogrel | Arm: Active Comparator: Control-ticagrelor
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/23 | 0/26
Serious Adverse Events (participants affected / at risk) | 1/25 | 0/23 | 0/26
Other Adverse Events (participants affected / at risk) | 14/25 | 11/23 | 13/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: CKD-Ticagrelor (N=25) | Arm: Active Comparator: CKD-Clopidogrel (N=23) | Arm: Active Comparator: Control-ticagrelor (N=26)
Hospitalization (Blood and lymphatic system disorders) | 1 (1) | 0 | 0 — for anemia requiring blood transfusion, possibly arising from worsening anemia of chronic kidney disease, no evidence of bleeding
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental: CKD-Ticagrelor (N=25) | Arm: Active Comparator: CKD-Clopidogrel (N=23) | Arm: Active Comparator: Control-ticagrelor (N=26)
Bruise (Injury, poisoning and procedural complications) | 12 | 9 | 13
Dyspnea (Cardiac disorders) | 5 | 1 | 1
Fatigue (General disorders) | 2 | 4 | 0
Acidity (Gastrointestinal disorders) | 0 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-02-22): https://cdn.clinicaltrials.gov/large-docs/11/NCT03649711/Prot_SAP_002.pdf
  • Informed Consent Form (2020-07-23): https://cdn.clinicaltrials.gov/large-docs/11/NCT03649711/ICF_003.pdf